CLINICAL TRIAL: NCT06980857
Title: Examining the Effect of the Physiotherapy Program Added to the ERAS Protocol on Pain, Function and Patient Satisfaction in Patients With Total Knee Arthroplasty
Brief Title: The Effect of the Physiotherapy Program Added to the ERAS Protocol in Patients With Total Knee Arthroplasty
Acronym: ERAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3/2022.K-86
Record Dates: First submitted 2025-02-03; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-02

CONDITIONS: Osteoartrit; ERAS protokolü; Total Diz Artroplastisi
Keywords: ERAS protokolü; Total diz artroplastisi
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Lower extremity exercises
  Interventions: Other: Control Group
- Eras Group (Active Comparator): Lower extremity exercises and early mobilization
  Interventions: Other: ERAS Group
- Multimodal physiotherapy group combined with ERAS protocol (Experimental): Preoperative pain education and home exercise brochure, early postoperative mobilization, lower extremity exercises, NMES current connection to quadriceps muscles in preop and postop process
  Interventions: Other: Multimodal physiotherapy group combined with ERAS protocol

INTERVENTIONS:
Other: Control Group — In our study, this group will be placed in hyperextension position and immobilized on postoperative day 0. Postop 1-2. Foot pumping exercises, isometric quadriceps exercises, passive knee extension, straight leg raising, 0-40 degree passive knee flexion, partial/full weight ambulation, respiratory exercises and cold application will be performed daily. On postoperative days 3-6 (depending on discharge time), stretching in passive knee extension, active/assisted quadriceps exercises, isometric-isotonic exercise for leg and hip muscles, 90-0 knee extension, 0-90 degree passive knee flexion exercises will be performed.
  Arms: control group
Other: ERAS Group — In our study, this group of patients were informed about the surgical procedure to be performed by the orthopedist; detailed information about the postoperative rehabilitation process, prevention of possible complications, preoperative nutrition, smoking and alcohol cessation time will be given. The patient will stop eating solid food 6 hours before the operation and stop drinking fluids 2 hours before the operation. Necessary consultations will be completed before surgery. Preoperative preparation of the patient will be organized according to the ERAS protocol. The patient will be mobilized early, either in bed or in the room, within 6-7 hours after surgery. The exercises of the first group will be continued from the first postoperative day.
  Arms: Eras Group
Other: Multimodal physiotherapy group combined with ERAS protocol — In our study, this group of patients who were informed about the surgery by the orthopedist will be examined by the anesthesiologist 1 week before surgery. Patients whose anesthesia preparation is completed will participate in a training program about pain, prevention of postoperative complications, auxiliary devices/equipment and exercises to be used, accompanied by a physiotherapist and a nurse. At the end of the program, patients will be given a 1-week home exercise program prepared by the physiotherapist. NMES device will be connected to the quadriceps muscles for 20 minutes half an hour before surgery, immediately after surgery and every day during hospitalization. Postoperatively, the patient will be mobilized early within 6-7 hours and the knee will be placed in hyperextension position. From the 1st day onwards, the exercises of the first group will be continued.
  Arms: Multimodal physiotherapy group combined with ERAS protocol

SUMMARY:
The aim of the study was to investigate the effects of bilateral total knee arthroplasty in patients with primary gonarthrosis ERAS protocol compared to standard rehabilitation protocol in the perioperative period to evaluate patients' pain, functional status and satisfaction. The main questions it aims to answer are:

* Physiotherapy applications added to the ERAS protocol after total knee arthroplasty are not effective on pain, function and patient satisfaction.
* Physiotherapy applications added to the ERAS protocol after total knee arthroplasty are effective on pain, function and patient satisfaction.

The investigators will be divided and allocated into 3 groups. Group 1 received standard treatment after TKA program will be applied, Group 2 will receive treatment with the ERAS protocol, and Group 3 will add a multimodal physiotherapy program to the ERAS protocol.

DETAILED DESCRIPTION:
After total knee arthroplasty (TKA), the patient must receive physical therapy to regain muscle strength, independent movement, and return to activities of daily living (ADL). One of the groups most frequently treated for rehabilitation during post-surgical hospitalization is patients who have undergone total knee arthroplasty surgery. Studies show that post-surgical patients return to their normal daily lives within approximately 6 weeks.However, complications, infections, limitation of the knee joint, additional post-surgical disorders, circulatory problems, vascular nerve problems, pain, rheumatic diseases affect the success of the surgery and the patient's recovery process.

Enhanced Postoperative Recovery Protocols (ERAS) are defined as a multidisciplinary approach that uses a combination of evidence-based practices to improve patient care. The treatment methods included in ERAS protocols are based on the understanding that the healing process can be optimized by protecting patients from catabolism and immune system disorders with factors such as pain management, regulation of fluid therapy, early mobilization and improvement of nutrition.This protocol includes a surgeon, anesthesiologist, nurse, dietitian and physiotherapist. The ERAS protocol considers the patient who will undergo surgery in 3 periods: preoperative period, intraoperative period and postoperative period. Starting with informing the patient before the surgery, bowel preparation, fasting period, alcohol and smoking cessation period, pre-surgical exercise training, surgical method, use of drains or tubes, type of anesthesia, post-surgical fluid intake, switching to carbohydrates, use of analgesia, early removal of tubes and drains. It covers principles such as removal and early mobilization. Looking at the results of research conducted by different disciplines, it is seen that the hospitalization period of patients applied to the ERAS protocol is shortened, their readmissions are reduced and complications are prevented.

Physiotherapy has a very small place in this multidisciplinary team. While it is mentioned that early mobilization plays a key role, it is not emphasized that exercise will accelerate mobilization, increase muscle strength and reduce pain.

Since the place of physiotherapy in the ERAS studies examined in the literature is limited and not comprehensive, the aim of this study is to evaluate the pain, function and patient satisfaction of the pre-op patient education, pain education, exercise, quadriceps muscle stimulation, post-op physiotherapy program applied in addition to the ERAS protocol in patients undergoing total knee arthroplasty. To investigate its effect on

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 60-80,
* Diagnosed with primary gonarthrosis,
* Individuals who decided to undergo total knee arthroplasty were included in the study.

Exclusion Criteria:

* Those with any neurological disease,
* Received physical therapy in the last 3 months,
* Those with cardiac problems (pacemarker),
* Those with systemic disease,
* Individuals who had revision surgery were not included in the study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 15 days
  A visual analog scale will be used to measure pain intensity and to monitor pain. This scale is a simple way to measure the intensity of pain. On a 10 cm horizontal scale, '0' means no pain and '10' means the most severe pain. A higher score indicates a worse outcome.
Oxford Knee Score | 15 days
  It will be used to assess physical function and pain. The Oxford Knee Score (OKS) developed by Dawson et al. is a 12-question reliable and validated questionnaire designed to assess pain and physical function based on the last 4 weeks in patients undergoing total knee arthroplasty. For each question, there are 5 response categories graded from 0 (worst) to 4 (best) points. Scores between 0-19 indicate severe knee arthritis, scores between 20-29 indicate moderate joint function, scores between 30-39 indicate mild joint function and scores between 40-48 indicate normal joint function. Items include pain, movement, limitation, standing up from a sitting position, squatting, walking up and down stairs, sleeping, housework, shopping, personal needs and transportation.
Hospital for Special Surgery | 15 days
  It will be used to assess pain, function, range of motion, muscle strength, deformity and instability in patients with total knee arthroplasty. It includes both objective and subjective assessment. The evaluation is based on 100 points. A score of 85 and above is considered excellent, 70-84 is considered good, 60-69 is considered fair and 60 and below is considered poor. A high score means that the results are good.
Timed Up and Go Test | 15 days
  It is done to measure the risk of falling and balance. The test requires a chair, a stopwatch and a 3-meter space. It is an easy test to perform with minimal equipment. The test measures the time between standing up from a sitting chair, walking 3 meters forward at normal speed, turning, walking 3 meters again, and sitting back in the chair. If a person completes this test in more than 12 seconds, they are at risk of falling. A longer duration means a poor outcome
Stair Climbing Test | 15 days
  A stair climbing test will be performed to assess lower limb strength, stair climbing ability and balance. Participants were asked to climb 9 steps with step intervals between 16-20 cm and the interval was recorded in seconds. A longer time means a poor result.
Assessment of Normal Range of Joint Motion | 15 days
  Normal range of motion and knee flexion-extension values will be assessed using a universal goniometer. During the measurement, the pivot point was taken as the lateral condyle of the femur and the fixed arm was placed parallel to the lateral midline of the femur. The mobile arm was positioned to follow the fibula. Goniometry is a simple instrument, easy to use and carry. It offers objective evaluation. In addition to assessing NEH, it is also used to determine a treatment program and to determine functional capacity.
Notthingam Health Profile | 15 days
  The Nottingham Health Profile will be used in our quality of life assessment. In the questionnaire consisting of 38 items, 6 different parameters related to health status are evaluated. These parameters are physical activity (8 items), emotional reactions (9 items), energy (3 items), social isolation (5 items), pain (8 items), and sleep (5 items). Each subparameter is scored between 0-100. A high score indicates worsening health. The total score is obtained by summing all sub-parameter scores.
Patient Satisfaction Survey | 15 days
  Participants' satisfaction will be evaluated with this scale After total knee arthroplasty (TKA), participants were asked whether they were satisfied with the surgical procedure. Patients were asked to rate their level of satisfaction on a scale of 1 to 5. Responses ranged from 1 - not at all satisfied to 5 - very satisfied. A high score means a high level of satisfaction. Participants' responses were recorded on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gül D Yılmaz Yelvar, Prof, Principal Investigator — Istinye University
Locations (1):
- İstinye Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No